CLINICAL TRIAL: NCT03876496
Title: A Phase One Feasibility Study of the Sensable®Care System: Establishing a Communications System for Patient Fall Reduction
Brief Title: Sensable®Care System: Establishing a Communications System for Patient Fall Reduction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: MedicusTek USA Corporation (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Kaiser Downey CTA
Record Dates: First submitted 2018-08-22; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Fall From Bed
Keywords: fall prevention; bed fall; acute care; patient safety; patient monitoring; health technology assessment; sensor devices and platforms; nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SensableCareCare System (Experimental): The Sensable®Care System uses pressure sensors and computer software to sense how patients are positioned on the bed in order to reduce bed falls. The Sensable®Care System Mattress has sensors embedded in them, which will be monitored by the nurses in the unit.
  Interventions: Device: SensableCare System

INTERVENTIONS:
Device: SensableCare System — The Sensable®Care Mattress has sensors embedded in it. Sensable®Care System is able to identify if the subject is stirring in bed, sitting up from the bed, attempting to leave the bed, or being out of the bed. If the subject is found to be in any of these four scenarios, four different types of alerts/notifications will warn clinicians: Stirring Notification, Sitting Up Notification, Bed Leaving Alert, Out of Bed Alert, will be generated by Sensable®Care System respectively.
  Once these four alerts/notifications are generated, designated attending nurses or caregivers equipped with a mobile app will receive audible, vibratory, and/or visual alerts from the Dashboard with subject's room number and type of alert displayed mobile app. Thus, interventions/assistance can be carried out presumably early. Harm to patient safety may be prevented.
  Other Names: MedicusTek

SUMMARY:
The purpose of this study is to test the effectiveness, safety and side effects of Sensable®Care System for inpatients. The Sensable®Care System uses pressure sensors and computer software to sense how patients are positioned on the bed in order to reduce bed falls. The Sensable®Care System Mattress has sensors embedded in them, which will be monitored by the nurses in your unit.

This study has three specific aims:

1. To assess the comfort of the system when used with hospitalized patients;
2. To observe how the system can be integrated into nurses' and hospital staff's regular workflow to help to modify and improve the system.
3. To analyze data from nursing response to alerts generated from hospitalized patients to improve alert system performance.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female
* Age: 18 years and older
* Racial and ethnic origin: all ethnic groups
* Hospital status: admitted in-patient or a patient under observation
* Expected hospital length of stay: minimum of 23 hours
* Willingness to participate in the study
* Moderate to High fall risk scoring a 2 or greater on the Mobility or Mental/LOC/Awareness status sections of the Hester Davis Fall Risk Assessment.

Exclusion Criteria:

* Declined to participate
* Patients less than 18 years old
* Patients who have been identified as a low fall risk or moderate fall risk with score less than 2 on the Mobility or Mental/ LOC/Awareness status sections of the Hester Davis Fall Risk Assessment
* Women who are documented as pregnant during the study period
* Patients who are medically unstable; as per the discretion of the primary nurse
* Patients who are actively in the dying process, at the discretion of the primary nurse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-09-24 (Actual); Primary Completion 2017-10-21 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
% of Nursing Staff Who Want to Use the System Following the Trial | focus group at week 8 within the 13 week study period
  Acceptance of SensableCare System after Trial Period
% of Nursing Staff Who Want to Use the System Following the Trial | focus group at week 12 within the 13 week study period
  Acceptance of SensableCare System after Trial Period

SECONDARY OUTCOMES:
Rate of Bed Falls Decreased Over Study Period | through the 13 week study period
  Whether bed falls had decreased over the study period compared to before the start of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Spicer, Principal Investigator — Kaiser Permanente
Locations (1):
- Downey Medical Center, Downey, California, United States